CLINICAL TRIAL: NCT01831882
Title: Identifying Biological Markers for Severe Depression
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Cornell University (Other); University of California, Irvine (Other); Pritzker Consortium (Other)
Responsible Party: Principal Investigator, Alan Schatzberg, Principle Investigator, Stanford University
Other Study IDs: 26529
Record Dates: First submitted 2013-04-09; First posted 2013-04-15 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will be retaining biospecimens including, whole blood, serum, hair and saliva tissues samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Major Depressive Disorder
- Healthy Control

SUMMARY:
The primary objective of this study is to investigate the biological components of major depression. The investigators are particularity interested in genetic variation and how it contributes to cortisol (because cortisol is higher in severe depression than mild depression or healthy controls) and how it contributes to clinical symptoms, especially suicidal ideation/behavior and psychosis.

ELIGIBILITY:
Inclusion criteria for depressed patients:

1. Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-IV) diagnosis of Unipolar Major Depressive Disorder with or without psychotic features.
2. 21-item Hamilton Depression Rating Scale (HDRS) score greater than or equal to 21.
3. Thase Core Endogenomorphic Scale score greater than or equal to 8 on the items included in the 21-item HDRS.
4. Between 18 - 70 years of age.
5. If currently taking antipsychotic, antidepressant, anticonvulsant, and/or mood-stabilizing medications, must be stable on the medication for at least one-week prior to entering the study.
6. Pre-existing (current) primary treating psychiatrist for subjects with psychotic features.
7. Any secondary diagnoses from the anxiety disorder spectrum is acceptable. Primary pre-existing chronic Obsessive-Compulsive Disorder (OCD) will be an exclusion criteria.

Inclusion criteria for healthy controls:

1. Between 18 - 70 years of age.
2. Have a HAM-D score of less than or equal to 5.

Exclusion Criteria for depressed patients:

1. Electroconvulsive Therapy (ECT) in the 6 months prior to the study.
2. Abuse of drugs or alcohol in the 6 months prior to study.
3. Unstable or untreated hypertension or cardiovascular disease.
4. Use of additional prescription medications, street drugs, or alcohol during the week before the study.
5. Any Axis II diagnosis or traits which would make participation in the study difficult.
6. Current pregnancy or lactation.
7. Post-partum depression
8. Diagnosis of obsessive-compulsive disorder
9. History of significant cognitive decline

Exclusion criteria for healthy controls:

1. Personal history of Axis I or Axis II disorders.
2. Active unstable medical problems.
3. Abuse of drugs or alcohol in the 6 months prior to study.
4. Use of additional prescription medications, street drugs, or alcohol during the week before the study.
5. Currently pregnant or lactating.
6. History of significant cognitive decline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatient hospitals, outpatient clinics, community.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Genetics | 1 year
  Blood will be drawn for gene expression, which includes genetics and metallothionein assessments. Blood will also be drawn for later assay of immune function/measures and neurotophins, and for future studies.

OTHER OUTCOMES:
Physiologic | 1 year
  Cortisol hormone levels will be measured in blood (suppression test), hair and saliva samples.
Neurocognition | 1 year
  Standardized neuropsychological measures will be used to assess neurocognition including, tests involving verbal learning, visual reproduction, attentional flexibility, and memory.
Clinical | 1 year
  Clinical psychiatric measures will be used to assess depression (HAM-D), psychotic features, suicidality, childhood trauma, and anhedonia.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Schatzberg, M.D., Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - University of California, Irvine, Irvine, California
  - Stanford University, Department of Psychiatry and Behavioral Sciences, Stanford, California
  - Weill Cornell Medical College, New York, New York